CLINICAL TRIAL: NCT00529932
Title: A Multi-Centre, Double-Blind, Randomised, Placebo-Controlled Trial Using CD133 Enriched Bone Marrow Cells Following Primary Angioplasty for Acute Myocardial Infarction
Brief Title: A Trial Using CD133 Enriched Bone Marrow Cells Following Primary Angioplasty for Acute Myocardial Infarction
Acronym: SELECT-AMI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Jozef Bartunek (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor-Investigator, Jozef Bartunek, Jozef Bartunek, Onze Lieve Vrouw Hospital
Organization: Onze Lieve Vrouw Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SELECT-AMI
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; Celltherapy; Bone Marrow

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Enriched CD133+, bone marrow-derived, autologous progenitor cells for this trial will be infused in the coronary arteries
  Interventions: Other: CD133+ infusion
- 2 (Placebo Comparator): Control group patients will receive 3 injections of 0.3 mL each of buffered normal saline (the vehicle used for cell suspension) into comparable vessels. Subjects will have an identical intra-coronary injection procedure to those randomized to autologous CD133+ progenitor cell injections.
  Interventions: Other: placebo infusion

INTERVENTIONS:
Other: CD133+ infusion — Subjects will be infused with all available autologous CD133+ cells after processing during one infusion session (during angiography).
  Arms: 1
Other: placebo infusion — Buffered normal saline will be infused in the coronary artery during an angiography.
  Arms: 2

SUMMARY:
An international, multi-centre, double-blind, randomised, placebo-controlled clinical trial with central core lab analyses to determine the safety of intra-coronary infusion of enriched CD133+, bone marrow-derived, autologous progenitor cells in patients 5-10 days after acute percutaneous coronary revascularization (primary PCI) for ST-segment elevation myocardial infarction (STEMI).

ELIGIBILITY:
Inclusion Criteria:

* Primary PCI for acute STEMI between 2-24 hours after onset of chest pain.
* ST-segment elevation >=2mm in >=3 adjacent leads.
* Presence of severe hypokinesia and/or akinesia in >=2 adjacent segments on echocardiogram at 48-72 hrs after primary PCI.
* Age between 20 and 75 years.

Exclusion Criteria:

* Pregnant or lactating.
* Prior history of myocardial infarction before index event.
* Decompensated congestive heart failure.
* Pre-existent LV dysfunction (EF <45% prior to admission)
* Cardiomyopathy.
* Previous cardiac surgery.
* Congenital heart disorder.
* Serum creatinine >200 Mmol/L.
* Presence of permanent pacemaker or implantable defibrillator.
* Contraindication to bone marrow aspiration.
* History of malignancy within 5 years except curatively treated basal cell carcinoma, squamous cell carcinoma and/or cervical carcinoma.
* Sustained or inducible VT >48 hours post primary PCI.
* Three vessel coronary artery disease necessitating intervention within 4 months.
* Immune compromise including chronic human immunodeficiency virus (HIV), hepatitis B virus (HBV) and hepatitis C virus (HCV) infection.
* Presence of chronic systemic inflammatory disorders.
* Previous autologous or allogeneic bone marrow or peripheral stem cell transplant or prior solid organ transplantation.
* Low hemoglobin, white blood cell, absolute neutrophil and/or platelet count.
* Any condition associated with a life expectancy of less than 6 months.
* Participation in unrelated research involving investigational pharmacological agent(s) 30 days before planned dosing.
* Current alcohol or drug abuse.
* Inability to provide written informed consent.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-09; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
PRIMARY SAFETY ENDPOINT Comparison of progression in coronary atherosclerosis burden proximal and distal to the stented segment of the infarct-related artery in treated and control groups. | at 6 months post-infusion
PRIMARY EFFICACY ENDPOINT Comparison of changes in myocardial thickening in non-viable akinetic / hypokinetic LV wall segments as determined by cardiac magnetic resonance imaging (cMRI) in treated and control groups. | at 6 and 24 months

SECONDARY OUTCOMES:
SECONDARY SAFETY ENDPOINT (a) Development of ventricular arrhythmias including failed sudden cardiac death. (b) Development of congestive heart failure. | At all follow up's
SECONDARY EFFICACY ENDPOINTS (a) Changes in % global LV ejection fraction (EF) compared with baseline as determined by cMRI and echocardiography pre- and post-cell infusion subsequent to primary PCI. | at all follow up's
SECONDARY EFFICACY ENDPOINTS (b)Assessment of epicardial resistance and microvascular resistance, index of myocardial resistance and absolute coronary blood flow measurements in the infarct related artery. | at 6 months follow up
SECONDARY EFFICACY ENDPOINTS (c) The feasibility of the CliniMACS® Reagent System to yield 5x106 CD133+ cells from 100-150 ml of autologous bone marrow. | prior to the infusion

CONTACTS AND LOCATIONS:
Overall Officials: Jozef Bartunek, MD, Study Chair — OLVZ Aalst; Jonathan Hill, MD, Study Chair — King's College London
Locations (5):
- Belgium (2):
  - OLVZ Aalst, Aalst
  - CHU ST-Pierre, Brussels
- Hôpital Cardiologique, Lille, France
- Catharina Ziekenhuis, Eindhoven, Netherlands
- King's College University Hospital, London, United Kingdom